CLINICAL TRIAL: NCT05247827
Title: The Effects of Targeted Phantom Motor Execution, Prosthetic Embodiment, and Surgical Closure on Phantom Limb Control, and Physical Function in People With Unilateral (Single) Transtibial (Below-the-knee) Amputation
Brief Title: The Effects of Targeted Phantom Motor Execution on Phantom Limb Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Audrey Zucker-Levin, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio 2855
Record Dates: First submitted 2022-01-25; First posted 2022-02-21 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Phantom Limb; Motor Activity; Amputation Stump; Amputation
Keywords: Prosthetic embodiment; Surgical closure; Phantom limb control; Physical function
MeSH Terms: conditions — Phantom Limb; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will receive usual and customary post-amputation treatment
- Exercise Group (Experimental): Participants will be trained for 3 consecutive weeks to perform the targeted exercise of their phantom limb in addition to receiving usual and customary post-amputation treatment.
  Interventions: Other: Targeted phantom limb motor execution (exercise)

INTERVENTIONS:
Other: Targeted phantom limb motor execution (exercise) — The targeted phantom motor execution is a specific training program for people with TTA that has been designed to improve the muscles' strength, coordination, and flexibility at the amputated and contralateral intact sides. Such training consists of repeated short-term, short rest interval, and moderate-intensity exercises (Schoenfeld 2010, Krutki, Mrowczynski et al. 2017). Targeted phantom motor execution can improve the body image considering its induced muscular impacts. People with TTA will be trained to follow specific movements of their foot-ankle complexes simultaneously, in order to increase PLA, as well as induce muscular morphologic and brain neuroplastic changes (Moseley and Brugger 2009).
  Arms: Exercise Group

SUMMARY:
Lower limb amputations account for more than 85% of all amputations. In Canada, it has been reported that transtibial amputation (TTA) is the most common level of amputation. Many people with limb amputation have awareness and feel that their missing limb still exists (phantom limb), with perceptions of sensation or pain, and the ability to move the limb with or without intention. Phantom limb sensation (PLS) is defined as all non-painful somatic sensations (e.g. sense of the limb position, touch, pressure, warmth or cold, or movement) in the missing part of the limb. The incidence of PLS is about 60% in adults after 17 months. In addition to PLS, 60-70% of people with amputation experience phantom limb pain (PLP), an intense chronic pain perception in their phantom limb, in the first year after amputation. Although PLP is well known to decrease the quality of life and lessen function, little is known about PLS and phantom limb control (PLC), the ability to intentionally move or control movements of the phantom limb. Enhancing PLS and PLC especially in the immediate months after amputation, could decrease painful perception, facilitate prosthetic control, and improve the function of people with amputations. Keeping this therapeutic and rehabilitative significance in mind, it is hypothesized that a targeted program of phantom motor execution, designed to address phantom limb awareness (PLA), the general knowledge of the presence or existence of the missing limb as one's own, could be associated with improving PLC in people with TTA. Furthermore, prosthetic embodiment, the sense that the prosthesis is accepted as a part of the body with the same functional abilities, may play a role in PLC. Investigating the association of PLC, as one of the phantom phenomena (i.e. PLA, PLS, PLP, and PLC), with surgical, clinical, and demographic characteristics of people with TTA will provide better insight into how phantom phenomena develop. The association of PLC with physical function has significant clinical importance that has never been investigated in people with TTA.

DETAILED DESCRIPTION:
This research explores testing of the following hypotheses with four independent but interrelated studies:

Study #1:

In people with TTA, post-amputation exercises focus on strength, balance, flexibility, and endurance training of the residual limb and intact limb muscles. Phantom limb motor execution, the active movement of the amputated body part, is not usually encouraged until a patient complains of PLP with the hypothesis that this intervention could re-organize the motor cortex to pre-amputation neural network and function. It was shown that phantom motor execution promoted by mirror therapy, virtual reality, and augmented reality could be used as a non-invasive therapy to relieve PLP in people with limb amputation. However, it is not clear if training with phantom motor execution improves peripheral control over the phantom limb. Therefore, this study explores the effects of a targeted phantom motor execution program on PLC in people with unilateral TTA.

Specific aim: To determine if targeted phantom motor execution improves control of the phantom limb, as measured by EMG patterning, in people with unilateral TTA.

Research hypothesis: People with unilateral TTA will improve control of their phantom limb after completion of a targeted phantom motor execution program.

Study #2:

Prosthetic embodiment is a sense that people with limb amputation feel that their prosthesis is integrated into their body and acts like their limb before amputation. It has been shown that higher prosthesis embodiment is associated with less PLP with the thought that it reverses brain plasticity after amputation. It is not clear whether prosthetic embodiment has any effect on PLC. This study explores the potential association between prosthetic embodiment and PLC in people with unilateral TTA.

Specific aim: To determine if there is a correlation between prosthetic embodiment, as measured by the self-reported TAPES-R and PEmbS-LLA questionnaires, and PLC (self-report), in people with unilateral TTA.

Research hypothesis: There is a strong positive association between prosthetic embodiment and PLC in people with unilateral TTA.

Study #3:

Surgical closure of the dissected muscles of the residual limb has been shown to impact PLP in people with limb amputation. The two most common surgical closure techniques are myodesis connection of the dissected muscles to bone/periosteum, and myoplasty, the connection of the dissected muscles to antagonist muscles. Residual limb muscles activity and PLA could be influenced by the distal closure of the dissected muscles. However, there is a scarcity of evidence on how surgical closure impacts the PLC. This study explores the association of surgical closure with PLC by measuring the symmetry of EMG muscle activity between the amputated and intact sides in people with unilateral TTA.

Specific aim: To determine if PLC, as measured by the symmetry of EMG muscle activity, is influenced by the surgical closure technique of the dissected muscles.

Research hypothesis: People who undergo unilateral TTA and myodesis surgical closure of the dissected muscles will have better PLC, as measured by the symmetry of EMG muscle activity, than those who undergo unilateral TTA and myoplasty surgical closure of the dissected muscles.

Study #4:

The previous three studies investigate the effects of the targeted phantom motor execution, prosthetic embodiment, and surgical closure on PLC. In the literature, it has been shown that improvement of PLC has been correlated with decreased PLP, and reduced PLP is associated with better function in people with limb amputation. However, it is not clear whether PLC has an association with physical function in people with TTA.

Specific aim: To determine if there is a correlation between PLC (self-report) and physical function, as measured by the four-square step test (FSST), in people with unilateral TTA.

Research hypothesis: There is a strong positive association between PLC and physical function in people with unilateral TTA.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Amputation surgery in Manitoba
3. Amputation surgery at least 6 months ago
4. Unilateral TTA
5. Existence of mature and wound-free residual limb
6. Experience of walking with a prosthesis for at least five months
7. Having contralateral healthy foot with no wounds, ulcers, abrasions, or loss of toes
8. Ability to walk independently for two minutes with/without an assistive device
9. Presence of PLA
10. Ability to read, write, and understand instructions and questionnaires in English
11. Have the dexterity to use a computer, tablet, or smartphone and the ability to communicate through Zoom application.

Exclusion Criteria:

1. Existence of psychological or psychiatric conditions (e.g. depression or anxiety) that negatively impact daily life
2. Addiction to alcohol or drug
3. Any medical condition that might conceivably alter how a person perceives the body or their ability to execute movements
4. Inability to move the intact limb at the foot and ankle joints
5. Fluctuating doses of pain suppressing medications in the previous month
6. Receiving formal training on exercising phantom limb
7. Existence of severe pain that limits activity
8. Undergoing prosthetic adjustments (e.g. in socket fit, components, alignment) in the past five months or plan to have prosthetic adjustments over the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Phantom limb control as measured by EMG patterning | 1 year (March 2022 - March 2023)
  The ability to intentionally move or control movements of the phantom limb
Prosthetic embodiment as measured by "Trinity Amputation and Prosthesis Experience Scales-Revised (TAPES-R)" | 1 year (March 2022 - March 2023)
  The sense that people with limb amputation feel that their prosthesis is integrated to their body and acts like their limb before amputation
Prosthetic embodiment as measured by "Prosthesis Embodiment Scale for Lower Limb Amputees (PEmbS-LLA)" | 1 year (March 2022 - March 2023)
  The sense that people with limb amputation feel that their prosthesis is integrated to their body and acts like their limb before amputation
Time score for four-square step test (s) | 1 year (March 2022 - March 2023)
  The fastest time required to pass through a sequence of 4 squares without touching the two crossing sticks that make those 4 squares. Both feet must make contact with the floor in each square while the person is face forward during the entire test.

SECONDARY OUTCOMES:
Amplitude of electromyography (EMG) of the agonist and antagonist muscles's activity | 1 year (March 2022 - March 2023)
  The maximum voltage of the EMG signal during activity of the agonist and antagonist muscles (i.e. Tibialis anterior, and Medial and Lateral Gastrocnemius) during targeted phantom motor executions
Frequency of electromyography (EMG) of the agonist and antagonist muscles's activity | 1 year (March 2022 - March 2023)
  The rate of EMG signal oscillation during activity of the agonist and antagonist muscles (i.e. Tibialis anterior, and Medial and Lateral Gastrocnemius) during targeted phantom motor executions
Index of electromyography (EMG) co-activation of the agonist and antagonist muscles | 1 year (March 2022 - March 2023)
  The amount of closeness of the EMG signal frequency of the agonist muscles to that of the antagonist muscles (the rate of EMG frequency of the agonist to that of the antagonist muscles' activity) during targeted phantom motor executions
Foot plantar load (N) | 1 year (March 2022 - March 2023)
  The measured load under the heel, midfoot, and toes of the foot during targeted phantom motor execution when measured by Loadsol insoles

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Zucker-Levin, Professor, Principal Investigator — University of Saskatchewan
Locations (1):
- Winnipeg Prosthetics and Orthotics (WinPO) Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
In Saskatchewan and Manitoba, the Health Information Protection Act (HIPA) defines how the privacy of participants' personal health information must be maintained so that their privacy and confidentiality will be respected. No information that discloses participant identity will be released or published without the participant's specific consent to the disclosure. However, research records and medical records identifying participants may be inspected in the presence of the principal investigator by the University of Saskatchewan Research Ethics Board for the purpose of monitoring the research. However, no records, which identify a participant by name or initials, will be allowed to leave the principal investigator's office. The results of this study may be presented in a scientific meeting or published, but the participants' identities will not be disclosed.

REFERENCES:
- [Background] Bekrater-Bodmann R, Reinhard I, Diers M, Fuchs X, Flor H. Relationship of prosthesis ownership and phantom limb pain: results of a survey in 2383 limb amputees. Pain. 2021 Feb 1;162(2):630-640. doi: 10.1097/j.pain.0000000000002063. PMID 32868751
- [Background] Brodie EE, Whyte A, Niven CA. Analgesia through the looking-glass? A randomized controlled trial investigating the effect of viewing a 'virtual' limb upon phantom limb pain, sensation and movement. Eur J Pain. 2007 May;11(4):428-36. doi: 10.1016/j.ejpain.2006.06.002. Epub 2006 Jul 20. PMID 16857400
- [Background] Dijkstra PU, Geertzen JH, Stewart R, van der Schans CP. Phantom pain and risk factors: a multivariate analysis. J Pain Symptom Manage. 2002 Dec;24(6):578-85. doi: 10.1016/s0885-3924(02)00538-9. PMID 12551807
- [Background] Flor H, Nikolajsen L, Staehelin Jensen T. Phantom limb pain: a case of maladaptive CNS plasticity? Nat Rev Neurosci. 2006 Nov;7(11):873-81. doi: 10.1038/nrn1991. PMID 17053811
- [Background] Geertzen JHB, van der Schans SM, Jutte PC, Kraeima J, Otten E, Dekker R. Myodesis or myoplasty in trans-femoral amputations. What is the best option? An explorative study. Med Hypotheses. 2019 Mar;124:7-12. doi: 10.1016/j.mehy.2019.01.008. Epub 2019 Jan 16. No abstract available. PMID 30798921
- [Background] Hunter JP, Katz J, Davis KD. The effect of tactile and visual sensory inputs on phantom limb awareness. Brain. 2003 Mar;126(Pt 3):579-89. doi: 10.1093/brain/awg054. PMID 12566279
- [Background] Hunter JP, Katz J, Davis KD. Stability of phantom limb phenomena after upper limb amputation: a longitudinal study. Neuroscience. 2008 Oct 28;156(4):939-49. doi: 10.1016/j.neuroscience.2008.07.053. Epub 2008 Aug 3. PMID 18755249
- [Background] Imam B, Miller WC, Finlayson HC, Eng JJ, Jarus T. Incidence of lower limb amputation in Canada. Can J Public Health. 2017 Nov 9;108(4):e374-e380. doi: 10.17269/cjph.108.6093. PMID 29120308
- [Background] Kilteni K, Groten R, Slater M. The Sense of Embodiment in Virtual Reality. Presence: Teleoperators and Virtual Environments. 2012; 21(4): 373-387.
- [Background] Krutki P, Mrowczynski W, Baczyk M, Lochynski D, Celichowski J. Adaptations of motoneuron properties after weight-lifting training in rats. J Appl Physiol (1985). 2017 Sep 1;123(3):664-673. doi: 10.1152/japplphysiol.00121.2017. Epub 2017 Jun 8. PMID 28596267
- [Background] Marshall HM, Jensen MP, Ehde DM, Campbell KM. Pain site and impairment in individuals with amputation pain. Arch Phys Med Rehabil. 2002 Aug;83(8):1116-9. doi: 10.1053/apmr.2002.33121. PMID 12161833
- [Background] Matjacic Z, Burger H. Dynamic balance training during standing in people with trans-tibial amputation: a pilot study. Prosthet Orthot Int. 2003 Dec;27(3):214-20. doi: 10.1080/03093640308726684. PMID 14727702
- [Background] Montoya P, Larbig W, Grulke N, Flor H, Taub E, Birbaumer N. The relationship of phantom limb pain to other phantom limb phenomena in upper extremity amputees. Pain. 1997 Aug;72(1-2):87-93. doi: 10.1016/s0304-3959(97)00004-3. PMID 9272791
- [Background] Moseley GL, Brugger P. Interdependence of movement and anatomy persists when amputees learn a physiologically impossible movement of their phantom limb. Proc Natl Acad Sci U S A. 2009 Nov 3;106(44):18798-802. doi: 10.1073/pnas.0907151106. Epub 2009 Oct 26. PMID 19858475
- [Background] Ortiz-Catalan M, Guethmundsdottir RA, Kristoffersen MB, Zepeda-Echavarria A, Caine-Winterberger K, Kulbacka-Ortiz K, Widehammar C, Eriksson K, Stockselius A, Ragno C, Pihlar Z, Burger H, Hermansson L. Phantom motor execution facilitated by machine learning and augmented reality as treatment for phantom limb pain: a single group, clinical trial in patients with chronic intractable phantom limb pain. Lancet. 2016 Dec 10;388(10062):2885-2894. doi: 10.1016/S0140-6736(16)31598-7. Epub 2016 Dec 2. PMID 27916234
- [Background] Rudy TE, Lieber SJ, Boston JR, Gourley LM, Baysal E. Psychosocial predictors of physical performance in disabled individuals with chronic pain. Clin J Pain. 2003 Jan-Feb;19(1):18-30. doi: 10.1097/00002508-200301000-00003. PMID 12514453
- [Background] Schafer ZA, Perry JL, Vanicek N. A personalised exercise programme for individuals with lower limb amputation reduces falls and improves gait biomechanics: A block randomised controlled trial. Gait Posture. 2018 Jun;63:282-289. doi: 10.1016/j.gaitpost.2018.04.030. Epub 2018 Apr 30. PMID 29804023
- [Background] Schoenfeld BJ. The mechanisms of muscle hypertrophy and their application to resistance training. J Strength Cond Res. 2010 Oct;24(10):2857-72. doi: 10.1519/JSC.0b013e3181e840f3. PMID 20847704
- [Background] Sin EI, Thong SY, Poon KH. Incidence of phantom limb phenomena after lower limb amputations in a Singapore tertiary hospital. Singapore Med J. 2013 Feb;54(2):75-81. doi: 10.11622/smedj.2013028. PMID 23462830
- [Background] Srinivasan SS, Gutierrez-Arango S, Teng AC, Israel E, Song H, Bailey ZK, Carty MJ, Freed LE, Herr HM. Neural interfacing architecture enables enhanced motor control and residual limb functionality postamputation. Proc Natl Acad Sci U S A. 2021 Mar 2;118(9):e2019555118. doi: 10.1073/pnas.2019555118. PMID 33593940
- [Background] Stankevicius A, Wallwork SB, Summers SJ, Hordacre B, Stanton TR. Prevalence and incidence of phantom limb pain, phantom limb sensations and telescoping in amputees: A systematic rapid review. Eur J Pain. 2021 Jan;25(1):23-38. doi: 10.1002/ejp.1657. Epub 2020 Sep 28. PMID 32885523
- [Background] Trevelyan EG, Turner WA, Robinson N. Perceptions of phantom limb pain in lower limb amputees and its effect on quality of life: a qualitative study. Br J Pain. 2016 May;10(2):70-7. doi: 10.1177/2049463715590884. Epub 2015 Jun 23. PMID 27551416
- [Background] Yaghi K, Yaghi Y, McDonald AA, Yadegarfar G, Cecil E, Seidl J, Dubois E, Rawaf S, Majeed A. Diabetes or war? Incidence of and indications for limb amputation in Lebanon, 2007. East Mediterr Health J. 2012 Dec;18(12):1178-86. PMID 23301391

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT05247827/Prot_SAP_000.pdf